CLINICAL TRIAL: NCT02338726
Title: Pelvic Floor Symptoms and Quality of Life in Elderly Women - a Population-based Pilot Study
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Virpi Rantanen, MD, Turku University Hospital
Other Study IDs: T268/2014
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Incontinence; Quality of Life
Keywords: urinary incontinence; pelvic floor; quality of life; elderly women
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Gynecological examination — Comparison of questionnaires and gynecological examination

SUMMARY:
To assess pelvic floor symptoms and quality of life in elderly women.

DETAILED DESCRIPTION:
The aim is to assess pelvic floor symptoms and quality of life in elderly women. The study is conducted as population-based in 100-130 women at the age of 64-66 years. All study objects are examined gynecologically and with vaginal ultrasound. Subjective symptoms are evaluated with validated questionnaires concerning pelvic floor symptoms, sexual symptoms and quality of life. This is a pilot study before a larger scale population-based study.

ELIGIBILITY:
Inclusion Criteria:

* All women in one municipality aged 64-66 years who are willing to participate in the study.

Exclusion Criteria:

* Persons under guardianship or who does not understand the used questionnaires.

Ages: 64 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100-130 women aged 64-66 years in one single municipality
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Validity of questionnaires to find pelvic floor symptoms | An average of 4 weeks, from returning the questionnaires to gynecological examination

SECONDARY OUTCOMES:
Quality of life in elderly women | ◦Measures assessed at the time when questionnaires are filled in, one time point

CONTACTS AND LOCATIONS:
Overall Officials: Virpi Rantanen, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland